CLINICAL TRIAL: NCT05701826
Title: Dose Escalation Study on the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of HRS3797 After Intravenous Infusion Administration in Healthy Adults
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of HRS3797 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fujian Shengdi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRS3797-103
Record Dates: First submitted 2023-01-18; First posted 2023-01-27 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Skeletal Muscle Relaxation

STUDY DESIGN:
Intervention Model Description: HRS3797 for dose escalation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Treatment group A1 (Experimental): HRS3797 for injection
  Interventions: Drug: HRS3797
- Treatment group A2 (Experimental): HRS3797 for injection
  Interventions: Drug: HRS3797
- Treatment group B1 (Experimental): HRS3797 for injection
  Interventions: Drug: HRS3797
- Treatment group B2 (Experimental): HRS3797 for injection
  Interventions: Drug: HRS3797
- Treatment group C1 (Experimental): HRS3797 for injection
  Interventions: Drug: HRS3797
- Treatment group C2 (Experimental): HRS3797 for injection
  Interventions: Drug: HRS3797

INTERVENTIONS:
Drug: HRS3797 — HRS3797 for injection, low dose
  Arms: Treatment group A1; Treatment group A2
Drug: HRS3797 — HRS3797 for injection, medium dose
  Arms: Treatment group B1; Treatment group B2
Drug: HRS3797 — HRS3797 for injection, high dose
  Arms: Treatment group C1; Treatment group C2

SUMMARY:
This is a single-center, open-label, dose-escalation study to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of HRS3797 in Chinese adults. To evaluate the effect of IV infusion duration on the safety, tolerability, pharmacokinetics and pharmacodynamics of HRS3797. To explore the ED95 dosage of HRS3797 in Chinese adults.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female subjects aged 18 to 45 years;
2. Conform to the ASA I Physical Status Classification;
3. Male subjects weighed ≥ 50kg, female subjects weighed ≥ 45kg, and body mass index (BMI) was in the range of 19.0~26.0 kg/m2 (inclusive);
4. No pregnancy plan for the next 3 months and voluntary use of highly effective contraception during the trial;
5. Able and willing to provide a written informed consent.

Exclusion Criteria:

1. Subjects with any clinically serious disease, such as circulatory, endocrine, nervous, digestive, respiratory, hematological, immunological, psychiatric, or metabolic abnormalities, that may affect the pharmacokinetic characteristics or safety evaluation of the investigational drug as determined by the investigator;
2. Subjects with neuromuscular disease;
3. Subjects with a history of anatomic airway abnormalities;
4. Subjects with any known allergy history or specific allergic diseases (e.g., allergic asthma, urticaria, eczema, etc.);
5. Subjects who underwent major surgery within 3 months prior to screening;
6. Subjects who underwent surgery that could significantly affect the pharmacokinetic characteristics or safety evaluation of the investigational drug, or who planned to undergo surgery during the study period;
7. Subjects who received antihistamines or antidepressants within 3 months prior to screening;
8. Subjects who used any drug that inhibits or induces liver metabolism of drugs (e.g., inducers - barbiturates, carbamazepine, phenytoin, glucocorticoids, omeprazole; Inhibitors - SSRI antidepressants, cimetidine, diltiazem, macrolides, nitroimidazoles, sedatives and hypnotics, verapamil, fluoroquinolones, antihistamines) within 30 days prior to administration;
9. Subjects who had used any medication within 14 days prior to administration;
10. Subjects who took other investigational drugs or used investigational devices within 3 months prior to the screening, or who planned to participate in other clinical trials during the study period;
11. Subjects who donated blood or suffered massive blood loss of >= 400 mL (except for physiological blood loss in women), received blood transfusions or used blood products within 3 months prior to the study, or planned to donate blood during the study period or within 1 month after finishing the study;
12. Subjects who smoked more than 5 cigarettes per day on average within 3 months prior to the study, or who could not quit smoking during the study period;
13. Subjects had a history of alcohol abuse within 3 months prior to the study, i.e., an average of more than 14 units of alcohol per week;
14. Subjects who consumed excessive amounts of tea, coffee, and caffeinated beverages within 3 months prior to the study;
15. Subjects who consumed special diet (e.g., grapefruit, grapefruit juice or food/drink containing grapefruit juice, chocolate, tobacco, alcohol, caffeine, etc.) within 48 hours before administration;
16. Subjects who have special requirements for diet and cannot comply with a unified diet;
17. The results of various examinations during the screening period were judged by the research doctor to be clinically significant abnormal;
18. Subjects who have one or more positive test results for hepatitis B virus surface antigen, hepatitis C virus antibody, human immunodeficiency virus antibody, and Treponema pallidum antibody;
19. Women who are pregnant or have a positive pregnancy test, or during breast-feeding;
20. Subjects with positive alcohol expiratory test results;
21. Subjects with positive smoking test results;
22. Not suitable to be included in the study for other reasons as considered by investigators.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-06-02 (Actual); Study Completion 2023-06-02 (Actual)

PRIMARY OUTCOMES:
Maximum T1 Suppression | 0 minute to full neuromuscular recovery after administration
Time to Maximum T1 Suppression | 0 minute to full neuromuscular recovery after administration
The onset of neuromuscular block | 0 minute to full neuromuscular recovery after administration
The duration of neuromuscular block | 0 minute to full neuromuscular recovery after administration
The recovery rate of neuromuscular block | 0 minute to full neuromuscular recovery after administration
Pharmacokinetic parameter of HRS3797: Cmax | 0 minute to 1.5 hour after administration
Pharmacokinetic parameter of HRS3797: AUC0-t | 0 minute to 1.5 hour after administration
Pharmacokinetic parameter of HRS3797: AUC0-∞ | 0 minute to 1.5 hour after administration
Pharmacokinetic parameter of HRS3797: Tmax | 0 minute to 1.5 hour after administration
Pharmacokinetic parameter of HRS3797: t1/2z | 0 minute to 1.5 hour after administration
Pharmacokinetic parameter of HRS3797: CLz | 0 minute to 1.5 hour after administration
Pharmacokinetic parameter of HRS3797: Vz | 0 minute to 1.5 hour after administration
The change of plasma histamine concentration from baseline | 0 minute to 1 hour after administration
The incidence and severity of adverse events/serious adverse events | from ICF signing date to day 28

SECONDARY OUTCOMES:
The ED95 dosage | 0 minute to full neuromuscular recovery after administration

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided